CLINICAL TRIAL: NCT04472780
Title: Effect of Hyperbaric Oxygen Therapy (HBOT) in Children With Autism Spectrum Disorder (ASD)
Brief Title: Hyperbaric Oxygen Treatment in Autism Spectrum Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Administration of Military Health, Tunisia (Network)
Collaborators: Military Hospital of Tunis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Autism spectrum disorder
Record Dates: First submitted 2020-06-03; First posted 2020-07-15 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Child Autism
Keywords: ASD - HBOT -
MeSH Terms: conditions — Autistic Disorder | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBOT Group (Experimental): will benefit from HBOT
  Interventions: Device: Hyperbaric oxygen Therapy HBOT
- Control group (No Intervention): will benefit from the conventional treatment

INTERVENTIONS:
Device: Hyperbaric oxygen Therapy HBOT — HBOT therapy protocol: in an eight-seat hyperbaric chamber 40 sessions of HBOT duration: 1 hour rhythm: 5 sessions / week pressure: 1.7 ATA (7 meters) O2 concentration: 100%
  Arms: HBOT Group

SUMMARY:
Hyperbaric oxygen therapy (HBOT) is part of a multidisciplinary therapeutic management of infant autism including psychotherapy, drug treatment and other therapeutics (speech therapy, occupational therapy restrictive diet ...).

It has been postulated that children with autism may benefit from HBOT due to the potential increase in cerebral perfusion occurring during treatment.

In fact, inhaling oxygen above atmospheric pressure could cause an increase in the arterial partial pressure of oxygen, leading to increased oxygen supply to the brain. HBO may also have anti-inflammatory properties due to the reduction in pro-inflammatory cytokines (tumor necrosis factor -α, interferon-γ and interleukins1 and 6). In addition, HBOT could improve mitochondrial dysfunction effects, as well as upregulate the production of antioxidant enzymes.Thus, hyperbaric oxygen therapy could be tried among the therapeutic arsenal of adjuvant treatments for autism.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder characterized by difficulties in verbal and non-verbal communication and social interactions. People with ASD often exhibit difficult behaviors, including aggressiveness, temper tantrums, irritability, hyperactivity, inattention, impulsivity, self-harm ..

The increasing prevalence of autism spectrum disorders (approximately 1%) has increased the need for evidence-based treatment to lessen the impact of symptoms.

The ethiopathogenesis of ASD has so far been unclear. Current pathophysiological theories have demonstrated the presence of cerebral hypo-perfusion, neuro-inflammation, immune dysregulation and oxidative stress involved in the genesis of this disorder. Based on its anti-inflammatory effects and increased amount of dissolved oxygen, hyperbaric oxygen therapy has been tried as one of the therapeutic arsenals of adjuvant therapy for autism.

This is a randomized controlled study including nearly 80 patients with ASD who underwent clinical and neuropsychological evaluation before and after HBOT treatment as well as the dosage of the various biochemical and immunological markers. These markers will be assessed before and after the HBOT. Perfusion MRI would also be performed before and after HBO.

ELIGIBILITY:
Inclusion Criteria:

* All children aged 4 to 14 years who were followed in the child psychiatry unit during the study period and who were identified as having a diagnosis of ASD. This diagnosis was made by child psychiatrists experienced in autism using the DSM-5 criteria and the ADI and the Childhood Autism Rating Scale (CARS)

Criteria for non-inclusion :

* Children with hearing or visual impairments
* Children with unbalanced epilepsy
* Children with a contraindication to HBOT
* Dysfunction of the immune system

Exclusion criteria

-Child that havent completed entire protocol

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
clinical severity assesement | 03 months
  Evaluate the interest of hyperbaric oxygen therapy in the management of ASD using CARS (child autism rating scale)

SECONDARY OUTCOMES:
dosage of Inetreleukine 6 | 03 months
  Evaluate the effect of HBOT on pro-inflammatory cytokines by Immunoassays: IL6
dosage of TNFα | 03 months
  Evaluate the effect of HBOT on pro-inflammatory cytokines by Immunoassays: TNFα
Oxidatif stress profil | 03 months
  Evaluate the effect of HBOT on the level of oxidative stress BY Biochemical dosages: Total antioxidant status (SAT)
dosage of Glutathione peroxidase | 03 months
  Evaluate the effect of HBOT on the level of oxidative stress BY Biochemical dosages: Glutathione peroxidase

CONTACTS AND LOCATIONS:
Locations (1):
- HBOT Department Military Hospital, Tunis, Montfleury, Tunisia

IPD SHARING:
Plan to Share IPD: No